CLINICAL TRIAL: NCT05585229
Title: Standardized Natural Psilocybin-assisted Psychotherapy for Tapering of Opioid Medication in Patients With Chronic Pain: an Open-label Feasibility Study
Brief Title: Standardized Natural Psilocybin-assisted Psychotherapy for Tapering of Opioid Medication
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Etheridge Foundation (Unknown)
Responsible Party: Principal Investigator, W Francois Louw, Clinical Associate Professor, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PsilOps
Record Dates: First submitted 2022-10-14; First posted 2022-10-18 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Opioid Dependence; Chronic Pain
Keywords: Opioid Tapering; Psilocybin; Psychotherapy; Chronic Pain; Hallucinogens; Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders; Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Psilocybin-assisted Psychotherapy (Experimental): Participants will undergo a single-arm, 8-week therapeutic intervention using natural standardized psilocybin-assisted psychotherapy as a treatment for opioid tapering in chronic pain patients. Specifically, they will undergo one or two standardized natural psilocybin (PEX010) dosing sessions; 25mg at week 3 and 37.5mg at week 7.
  Interventions: Drug: Psilocybin-assisted Psychotherapy

INTERVENTIONS:
Drug: Psilocybin-assisted Psychotherapy — Participants will complete a 8-week structured psychotherapeutic intervention involving administration of 25mg and 37.5mg PEX010 on two separate occasions.
  Other Names: PEX010

SUMMARY:
This is an open-label pilot trial to assess the safety and feasibility of a novel 8-week psilocybin-assisted psychotherapy intervention to facilitate successful tapering/discontinuation of opioid pain medication in adult patients receiving long-term opioid therapy for chronic pain. Participation will last approximately 8 months and includes one or two psilocybin-assisted therapy sessions. The study will evaluate the incidence and severity of adverse events during and after treatment, the number of participants who drop out of the study for intervention-related reasons, and the self-reported benefits and harms of the intervention.

DETAILED DESCRIPTION:
The purpose of this pilot study is to establish the safety and tolerability of a therapeutic intervention using psilocybin-assisted psychotherapy as a novel treatment for opioid tapering in a sample of patients with chronic pain. Participants will be patients who have failed previous attempts to reduce their use of opioid medication and who have no medical or psychological contraindications for psilocybin administration.

This pilot study involves an 8-week open-label, non-randomized therapeutic intervention and a 6-month follow-up period. To provide a supportive context for the drug experience, participants will receive preparatory and integrative sessions following an acceptance and commitment therapy model for psychedelic therapy. The physician-supervised opioid taper will begin following the first psilocybin dosing session (25mg) after an integration session with therapists, and a second optional psilocybin dosing session (37.5mg) will be facilitated one month later. Assessments will be completed at baseline, and at follow-up points at 1-month, 3-months and 6-months post-intervention to evaluate both acute and long-term effects of the intervention.

Primary outcomes of interest are rates of adverse events, retention rates, and patient perceptions of intervention tolerability. Preliminary efficacy of the treatment will be evaluated by tracking opioid reduction rates and long-term maintenance of these reductions. Other measures of interest include qualities of the psychedelic experience, opioid cravings and withdrawal, chronic pain symptoms, and psychological mechanisms.

ELIGIBILITY:
Inclusion Criteria:

1. Must be 19 - 75 years of age.
2. Have a diagnosed noncancer chronic pain condition including but not limited to neuropathic pain, fibromyalgia, chronic headaches/migraines, back pain, musculoskeletal pain.
3. Currently on a stable dose of opioid therapy on short-acting, long-acting, or combination of opioid medication types, for a minimum duration of 90 consecutive days.
4. History of at least one unsuccessful attempt to taper or discontinue long-term opioid therapy, and has expressed current interest in making another attempt to reduce or discontinue.
5. Able to swallow capsules/tablets.
6. If of childbearing potential, agree to practice an effective means of birth control throughout the duration of the study.

Exclusion Criteria:

1. Have any of the following cardiovascular conditions: uncontrolled hypertension, coronary artery disease, congenital long QT syndrome, cardiac hypertrophy, greater than first degree AV block, cardiac ischemia, congestive heart failure, myocardial infarction, tachycardia, chronic bradycardia, artificial heart valve, a clinically significant screening ECG abnormality, or any other significant cardiovascular condition.
2. Asthma
3. Have moderate to severe hepatic impairment.
4. Chronic pain is due to cancer.
5. Women who are pregnant, who intend to become pregnant during the study, or who are currently breastfeeding.
6. Have a history of stroke or Transient Ischemic Attack (TIA).
7. Meet DSM-5 criteria for severe alcohol or drug use disorders (other than Opioid use Disorder).
8. Nicotine dependence that would prevent the participant from remaining nicotine free for the duration of dosing sessions (i.e., 6-8 hours).
9. Have Epilepsy.
10. Clinically significant sleep disorders such as sleep apnoea not on appropriate treatment.
11. Have Insulin-dependent diabetes.
12. Participants who are or have been taking mood stabilizers (e.g. lithium), SSRIs/SNRIs (e.g. citalopram, venlafaxine, vortioxetine, duloxetine), herbal remedies with serotonin activity (e.g. 5-HTP, St. John's Wort), dopamine agonists (e.g. bupropion), tricyclic antidepressants (e.g. amitriptyline), antipsychotics (e.g. haloperidol), amphetamines (e.g. amphetamine/dextroamphetamine salts, methylphenidate, dextroamphetamine, lisdexamfetamine), monoamine oxidase inhibitors (e.g. isocarboxazid, phenelzine, selegiline, tranylcypromine), alcohol or aldehyde dehydrogenase inhibitors (e.g. disulfiram), and UDG modulators (i.e. UGT modulators such as phenytoin, regorafenib, eltrombopag) during the study or in the preceding 8 weeks.
13. Hallucinogenic or psychedelic drug use within 12 months (i.e. any use of mescaline, 2C-B, psilocybin, LSD, 5-MeO-DMT, ibogaine ayahuasca, MDA, MDMA, ketamine or any related molecules).
14. Meet DSM-5 criteria for schizophrenia spectrum or other psychotic disorders, including major depressive disorder with psychotic features, or Bipolar I or Bipolar II Disorder.
15. Have a first degree relative with schizophrenia, Bipolar I or Bipolar II Disorder.
16. Meet DSM-5 criteria for diagnosis of antisocial or borderline personality disorders.
17. Participants with a history of a developmental disorder.
18. Participants diagnosed with serious comorbidities that may or may not influence mental health in the opinion of the qualified investigator.

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-10-27 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of psilocybin administration | Week 31
  Percentage of participants who provide consent and complete the intervention.
Acceptability of psilocybin administration | Week 31
  Participant ratings of benefits and harms of the intervention.
Safety of psilocybin administration | Up to 33 Weeks
  Number and type of treatment-related adverse events and serious adverse events reported during the intervention.

SECONDARY OUTCOMES:
Change in prescribed opioid dose at the 1-month visit compared to initial dose | Week 11
  Taper adherence rates will be assessed by categorizing participants as "adhering", or "non-adhering" based on percentage of the initial dose that they are using at the 1-month timepoint.
Change in prescribed opioid dose at the 3-month visit compared to initial dose | Week 19
  Taper adherence rates will be assessed by categorizing participants as "adhering", or "non-adhering" based on percentage of the initial dose that they are using at the 3-month timepoint.
Change in prescribed opioid dose at the 6-month visit compared to initial dose | Week 31
  At 6-month follow-up participants will be categorized as "successful" if they have discontinued opioid therapy, and "unsuccessful" if they have not.

CONTACTS AND LOCATIONS:
Overall Officials: W. Francois Louw, MD, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia - Okanagan Campus, Kelowna, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No